CLINICAL TRIAL: NCT03187444
Title: Cardiovascular Risk and Chronic Inflammatory Rheumatism
Acronym: RCVRIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHU-337; 2014-A01847-40 (Other: 2014-A01847-40)
Record Dates: First submitted 2017-06-07; First posted 2017-06-15 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2017-06

CONDITIONS: Rheumatology; Cardiovascular Diseases; Arthritis, Rheumatoid; Spondyloarthritis
Keywords: Cardiovascular risk; Chronic inflammatory rheumatism; Rheumatoid arthritis; Spondyloarthritis; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Arthritis, Rheumatoid; Spondylarthritis; Inflammation | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: all participants receive the same intervention throughout the protocol
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic inflammatory rheumatism (Experimental): All patients over 18 years, with rheumatoid arthritis treated for the first time with conventional anti-TNF therapy, Abatacept, Tocilizumab, Rituximab or patients with spondyloarthritis treated for the first time with NSAIDs that may be associated with conventional background treatments for peripheral or biological (anti-TNF, Usketinumab) may be included.
  Interventions: Procedure: Examinations

INTERVENTIONS:
Procedure: Examinations — Several examinations are realized on each patients, in addition to the usual visit and after verification of the criteria of inclusion and signature of consent.

SUMMARY:
Chronic inflammatory rheumatism and inflammation can increase the risk of cardiovascular problems. Indeed, these diseases can increase the risk of myocardial infarction. The objective of this project is a better understanding and preventing the risk of cardiovascular problems in chronic inflammatory rheumatism through the study on the long-term flexibility of the arteries, blood markers of cardiovascular risk and muscle mass.

DETAILED DESCRIPTION:
All patients over 18 years, with rheumatoid arthritis treated for the first time with conventional anti-TNF therapy, Abatacept, Tocilizumab, Rituximab or patients with spondyloarthritis treated for the first time with NSAIDs that may be associated with conventional background treatments for peripheral or biological (anti-TNF, Usketinumab) may be included. However, they must be subject to a Social Security scheme and will only be able to participate in the research if they give their consent in writing after receiving full information.

In addition to the usual visit and after verification of the criteria of inclusion and signature of consent, arterial stiffness and endothelial function measurement are performed at M0, M6, M12 and every year and also at each change of treatment, By measuring the pulse wave velocity and by determining the Alx by the SphygmoCor XCEL (AtCor Medical Pty Ltd, based in Australia (CE 0120). Cardiac Frequency at rest will be evaluated at M0, M6, M12, every year and also at each change of treatment, by the realization of an electrocardiogram. The intima-media thickness (EIM) of the carotid will be evaluated every 5 years According to the recommendation. EIM is a non-invasive ultrasound technique in which an ultrasound probe is placed opposite the right primitive carotid artery by convention. A measurement of endothelial function will be performed at M0, M6, M12 and then every year in patients

A study of regional myocardial function by high-resolution echocardiography-STI will be carried out at M0, M6, M12 and then every year in non-hypertensive patients, without diabetes, without a cardiovascular history.

A Serum / plasma / urine bank will be constituted at M0, M6, M12, every year and also at each change of treatment to determine the markers of cardiovascular risk. The plasma bank will be used for the determination of nitric oxide.

A study of the body composition dual-energy x-ray absorptiometry (DXA) and pQCT allowing to evaluate lean mass, fat mass and bone mineral mass will be carried out at M0, then every year and also at each change of treatment M6 assessment of lean mass and fat mass only). When DXA is examined, a lateral incidence measurement of the rachis will be performed to calculate an arterial calcification score.

Muscle strength will be measured by hydraulic hand dynamometer Jamar (Kinetec company) at M0, M6, M12 then every year and also at each change of treatment. Physical performances will be evaluated by a 6-minute walking test, 10 meters walking speed and "Timed up-and-go test" stool test, which combines both coordination mechanisms, proprioception and muscular strength of lower limbs than M0, M6, M12 and then every year and also with each change of treatment.

The physical activity and physical inactivity of the patient and food habits will be assessed by the GPAQ (Global Physical Activity Questionnaire), FFQ and a Food questionnaire to M0, M6, M12 and every year and also to each change of treatment .

Depression will be assessed by the HAD self-administered questionnaire at M0, M6, M12 and then every year and also at each change of treatment.

Fibromyalgia will be assessed by the Fibromyalgia Rapid Screening Tool at M0, M6, M12 and then annually.

Comorbidities will be assessed by a nurse at M0, M12 and then annually.

All these examinations will be carried out in addition to the usual follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years
* Have rheumatoid arthritis or spondyloarthritis (ankylosing spondylitis, psoriatic arthritis)
* Receive first conventional DMARD or biological treatment (anti-TNF, Abatacept, Tocilizumab, rituximab) for patients with rheumatoid arthritis
* Receive biological treatment (Abatacept, Tocilizumab, rituximab) for patients with rheumatoid arthritis who have failed anti-TNF treatment.
* Receive first NSAID (optionally combined with conventional DMARDs in case of peripheral arthritis) or biological treatment (anti-TNF, Usketinumab) for patients with spondyloarthritis.
* Being subject to a social security scheme
* Have the capacity to give informed consent and to comply with the study requirements

Exclusion Criteria:

* Patient refused to sign the consent form
* Patient under guardianship
* Patient having already been exposed to a biological as part of its pathology
* Patient with chronic disease may interfere with cardiovascular disease either by itself or by treatment history
* For echocardiography high resolution STI: Patients with hypertension, diabetes and cardiovascular history.
* To evaluate the activity of the autonomic nervous system, patients with hypertension, diabetics, with cardiovascular history with a neurological disease, with vasoactive or chronotropic treatments such as beta-blockers, antiarrhythmics, antihypertensives, anxiolytics, antidepressants
* Pregnant or lactating women will be temporarily excluded from the study during the period of pregnancy and breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-04-24 (Actual); Primary Completion 2036-10-24 (Estimated); Study Completion 2037-04-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the arterial Stiffness | at 6 months, 12 months
  evaluated by the pulse wave velocity
Change from baseline of resting heart rate | at 6 months, 12 months
Change from baseline of endothelial function | at 6 months, 12 months
  by Tonometry
Change from baseline of intima-media thickness and carotid and femoral atheroma | at 5 years
Change from baseline of autonomic nervous system activity | at 6 months, 12 months
Change from baseline of regional myocardial function | at 6 months, 12 months
Change from baseline of other markers of cardiovascular risk | at 6 months, 12 months
  troponin, NT_proBNP, adipocytokines, MCP-1, assymetric dimethylaarginine, angiopoietin-2, anti apo A-1, IL-6, IL-17
Change from baseline of an abdominal aortic calcification score (DEXA) | at 6 months, 12 months
Change from baseline of hand muscle strength (Handgrip) | at 6 months, 12 months
Change from baseline of energy expenditure and physical activity in usual living conditions | at 6 months, 12 months
  by Android application on smartphone (eMeetingSearch)
Change from baseline of food habits | at 6 months, 12 months
  French FFQ questionnaire
Change from baseline of body composition | at 6 months, 12 months
  DEXA, pQCT
Change from baseline of inflammatory rheumatism | at 6 months, 12 months
  by the doctor in charge of the patient
Change from baseline of depression (HAD) | at 6 months, 12 months
Change from baseline of fibromyalgia (FIRST) | at 6 months, 12 months
Change from baseline of the frequency of comorbidities during inflammatory rheumatism | at 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin SOUBRIER, PhD MD, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France